CLINICAL TRIAL: NCT00290550
Title: A Phase IIA Study Evaluating the Efficacy of MK0457 as a 5-Day Continuous Infusion in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Phase IIA Study of MK0457 in Patients With Cancer of the Lung (0457-006)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0457-006; 2006_008
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Advanced Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tozasertib

ARMS (1):
- 1 (Other): MK-0457
  Interventions: Drug: MK0457

INTERVENTIONS:
Drug: MK0457 — IV infusion at 10 mg/m2/hour; 5-day continuous infusion every 21 days

SUMMARY:
This is a study to evaluate the effectiveness of an investigational drug in patients with cancer of the lung.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age with cancer of the lung and who have had either no previous treatment or 1 previous treatment for advanced cancer of the lung. Certain other treatments may also be allowed (prior cytotoxic chemotherapy in the adjuvant setting)

Exclusion Criteria:

* Patients who have had treatment with any investigational therapy within the past 30 days are not eligible.
* Patients who have had a disease or medical condition that is not controlled will not be eligible.
* Patients who are pregnant or breastfeeding are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of MK0457 as a 5 day infusion as measured by radiological exams at baseline and after every other cycle of treatment. After 3 post-treatment radiological assessments, response will be measured after every third cycle. | 5 Days

SECONDARY OUTCOMES:
Safety and tolerability as measured by duration, intensity (grade) and time of onset of toxicity. | 5 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC